CLINICAL TRIAL: NCT06664164
Title: Comparison of Postoperative Analgesic Efficacy of Adjuvant Quadratus Lumborum Block in Open Technique Inguinal Hernia Surgeries
Brief Title: Postoperative Analgesic Efficacy of Adjuvant Quadratus Lumborum Block in Open Inguinal Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, principal investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GAZIAOSMANPASA TREHAQ
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative
Keywords: anterior quadratus lumborum block; postoperative pain; adjuvant; dexamethasone; inguinal hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Everyone except the person preparing the medication for the patient will be blinded. The person performing the block, the participants, and those monitoring during the postoperative period will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB Group (Active Comparator): anterior quadratus lumborum block group
  Interventions: Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK
- adjuvant QLB Group (Active Comparator): with adjuvant anterior quadratus lumborum block group
  Interventions: Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK WİTH ADJUVANT

INTERVENTIONS:
Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected.
  Arms: QLB Group
Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK WİTH ADJUVANT — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine and 8 mg de-xamethasone are injected.
  Arms: adjuvant QLB Group

SUMMARY:
Evaluation of Postoperative Analgesic Efficacy of Adjuvant Use in Quadratus Lumborum Blocks

DETAILED DESCRIPTION:
primary aim : Compare the time to first rescue analgesia in patients following the application of non-adjuvant Quadratus Lumborum Block and adjuvant Quadratus Lumborum Block for postoperative analgesia after inguinal hernia surgeries performed under spinal anesthesia.

secondary aims are to: to compare and evaluate the total analgesic consumption over 24 hours Compare NRS (Numerical Rating Scale) values (at rest and dynamic) in patients during postoperative follow-ups at 4, 8, 12, and 24 hours.

Compare side effects such as postoperative nausea and vomiting. In trunk blocks, local anesthesia is applied to the interfascial area between the abdominal wall or back muscles. Local anesthetics and steroids are used for this purpose. The analgesic efficacy of steroids is known from their perineural applications. Due to the lack of blood circulation and vascularization in the interfascial area, the absorption of local anesthetics is slow, providing prolonged analgesic effects. Trunk blocks applied in these regions are used as part of multimodal analgesia. The effectiveness of trunk blocks may vary based on the patient's anatomical differences and previous surgeries, but analgesic efficacy is generally observed for an average of 8-12 hours. the investigators believe that with the use of adjuvants, these durations will be extended, and analgesic efficacy will increase.

In this study, it is planned to add a total of 8 mg of dexamethasone to the local anesthetic agent for patients undergoing adjuvant anterior Quadratus Lumborum Block. In studies conducted in the field of trunk blocks, the expected duration of analgesia is an average of 8-12 hours. In this study, the block application is planned to be preoperative. Dexamethasone was chosen as an adjuvant to extend the expected analgesia duration of 8-12 hours and to increase analgesic efficacy. Dexamethasone is known to be effective and safe when used as an adjuvant in all nerve blocks.

To reduce opioid-related side effects such as nausea, vomiting, itching, constipation, and dependence associated with opioid medications used in postoperative analgesia for inguinal hernia surgeries, opioid-sparing analgesia and regional techniques are being employed. Quadratus Lumborum Blocks are being safely and easily performed and are frequently preferred in abdominal surgery due to recent advancements in trunk block techniques and ultrasound technology.

This study aims to evaluate the postoperative analgesic efficacy of adjuvant and non-adjuvant anterior Quadratus Lumborum Blocks in patients undergoing inguinal hernia surgery. The investigators predict that the analgesic efficacy of the adjuvant Quadratus Lumborum Block will be more effective and longer-lasting.

ELIGIBILITY:
Inclusion Criteria: - 18-65 years, American Society of Anesthesiologists physical statusⅠ-II -

Exclusion Criteria:

* local anesthetic allergy
* Infection at the procedure site
* Body Mass Index >35 kg/m2
* Anticoagulant use with bleeding disorder
* Chronic analgesia and opioid use -with mental and psychiatric disorders -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
time to first rescue analgesic requirement. | 24 hour
  Compare the time to first rescue analgesia in patients

SECONDARY OUTCOMES:
Total analgesic Consumption | 24 hour
  Our primary aim is to compare and evaluate the total analgesic consumption(diclofenac) over 24 hours following the application of non-adjuvant Quadratus Lumborum Block and adjuvant Quadratus Lumborum Block for postoperative analgesia after inguinal hernia surgeries performed under spinal anesthesia.
To compare the NRS (Numering rating scale) values (resting and dynamic) at 4. 8. 12 . 24. hours in the postoperative follow-up of the patients | 24 hour
  Compare NRS (Numerical Rating Scale) values (at rest and dynamic) in patients during . postoperative follow-ups at 4, 8, 12, and 24 hoursAssessed at various time points to quantify pain intensity at rest and during movement. The Numerical Rating Scale (NRS) is a pain assessment tool where patients rate their pain from 0 (no pain) to 10 (worst pain).
To compare postoperative side effects such as nausea, vomiting | 24 hour
  To compare postoperative side effects such as nausea, vomiting, quadriceps weakness

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Sehirlioglu, MD, Principal Investigator — Gaziosmanpasa Research and Training Hospital
Locations (1):
- Gaziosmanpasa Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: always
Access Criteria: drserpilsahin@gmail.com

REFERENCES:
- [Background] Priyadarshini K, Behera BK, Tripathy BB, Misra S. Ultrasound-guided transverse abdominis plane block, ilioinguinal/iliohypogastric nerve block, and quadratus lumborum block for elective open inguinal hernia repair in children: a randomized controlled trial. Reg Anesth Pain Med. 2022 Apr;47(4):217-221. doi: 10.1136/rapm-2021-103201. Epub 2022 Jan 17. PMID 35039439
- [Background] Favaro ML, Gabor S, Souza DBF, Araujo AA, Milani ALC, Ribeiro Junior MAF. Quadratus Lumborum Block As A Single Anesthetic Method For Laparoscopic Totally Extraperitoneal (Tep) Inguinal Hernia Repair: A Randomized Clinical Trial. Sci Rep. 2020 May 22;10(1):8526. doi: 10.1038/s41598-020-65604-x. PMID 32444629